CLINICAL TRIAL: NCT02382081
Title: A Randomized Control Trial of Patient-initiated Hospital Follow-up for Patients With Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Lina R. Khoury, B.N., stud.cand.scient.sant, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Behov
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient-initiated shared care (Experimental): Patient-initiated shared care hospital reviews in which there were one planed hospital review every year and if needed additional reviews initiated by the patient.
  Access to nurse-run telephone helpline with direct access to a contact nurse.
  Interventions: Procedure: Patient-initiated shared care
- Control (No Intervention): Traditional, routine hospital reviews every three-fourth month.

INTERVENTIONS:
Procedure: Patient-initiated shared care
  Arms: Patient-initiated shared care

SUMMARY:
The primary objective of this research protocol is to evaluate the health related quality of life and efficacy of patient-initiated hospital follow-up for patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease affecting 1 to 3% of the European population. Treatment of moderate to severe psoriasis often requires lifetime routine reviews by hospital dermatologist. Patterns of hospital review vary, but most patients attend follow-up every 12-16 week by dermatologist. At routine reviews the patient disease is often quiet and little intervention or no intervention is required, and times were the patient need help the time is limited for in-depth consultation. Both patient and healthcare professional requested more time. In-depth consultation is important in the care of psoriasis, because moderate to severe psoriasis has a significant impact on quality of life and patient have an increased incidence of cardiovascular risk factors such as hypertension, overweight, hyperlipidemia and exposure to tobacco and alcohol. These comorbidities and the psychosocial burden must be addressed by clinicians to help patients to acquire or to maintain competencies that are required to live with a chronic disease.

Patient-initiated hospital follow-up for patients with moderate to severe psoriasis might reduce inappropriate follow-up appointments, improve rapid access to specialist care and release resource to further in-depth consultation. If the patient is empowered to initiate hospital review thus patient's individual needs dictate the content, duration and contact with clinicians. It is our goal that an individual needs-based patient involvement in the shape of patient-initiated hospital follow-up,will be perceived as a benefit of the patients who 1) meets a high safety in the patient's own provision of medical treatment, 2) increase the patient's knowledge of the lifestyle and prevention of comorbidities and 3) strengths patient's overall satisfaction with treatment.

ELIGIBILITY:
Inclusion Criteria:

• Patients in stable systemic psoriasis treatment defined as having received treatment for more then 12 weeks without complication and being adherence to medication administration.

Exclusion Criteria:

* Patients not able to give informed consent
* Patients not able to follow the program
* Patient with server psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-05-02; Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Dermatology life quality index (DLQI) | 2 years
  Evaluation of quality of life

SECONDARY OUTCOMES:
SF36 - Short Form 36 (SF-36) | 2 years
Psoriasis Area and Severity Index (PASI | 2 years
Hospital Anxiety and Depression Scale (HADS) | 2 years
Body Image Scale (BIS) | 2 years
Self-developed patient safety scale | 2 years
Hospital visits | 2 years
Numbers of phone calls to the nurse-run telephone helpline | 2 years
Adherence to medicine treatment | 2 years
Charlson Comorbidity Index | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Khoury LR, Moller T, Zachariae C, Skov L. A prospective 52-week randomized controlled trial of patient-initiated care consultations for patients with psoriasis. Br J Dermatol. 2018 Aug;179(2):301-308. doi: 10.1111/bjd.16369. Epub 2018 May 23. PMID 29363093